CLINICAL TRIAL: NCT02677363
Title: Functional Outcomes of Stay Strong, Stay Healthy Program
Brief Title: Functional Outcomes of Stay Strong Stay Healthy Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 208531
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Quality of Life; Aging; Memory Loss; Cardiovascular Diseases
Keywords: Elderly; Older; Adults; Resistant Exercise; Strength Training; Cognitive function
MeSH Terms: conditions — Memory Disorders; Cardiovascular Diseases | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Older adults (Experimental): Participants 60 and above aged (both females and males) will perform one hour of resistance exercise twice weekly for 8 weeks.
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — Participants 60 and above aged (both females and males) will perform one hour of resistance exercise twice weekly for 8 weeks.
  Other Names: Strength training

SUMMARY:
Strength training can increase muscle mass and strength while improving bone density and reducing risk for osteoporosis and related fractures. Strength training can also lead to reduced risk for diabetes, heart disease, arthritis, depression, and obesity; and improves self-confidence, sleep and vitality. Research demonstrates that strength training is extremely effective in helping aging adults with chronic conditions prevent further onset of disease and, in many instances, actually reverse the disease process. In Stay Strong, Stay Healthy Program elderly subjects perform resistance exercise training (RET) twice every week. Past literature suggests that resistance training improved muscle activity, muscle strength, muscle mass, and bone mineral density and total body composition, and adiponectin, insulin sensitivity, fasting blood-glucose (BG), HbA1c1 (long-term marker of BG), blood pressure (BP), blood triglycerides (TGs) and low density lipoproteins (LDL) in healthy and diabetic subjects. The purpose of this study is to measure the changes in the above discussed variables after 8-weeks of resistance exercises.

DETAILED DESCRIPTION:
Participants will perform resistance exercise for 8 weeks and measurements (anthropometric, electromyography, pulse wave velocity, strength test, dual x-ray absorptiometry, blood enzymes/hormones, and sleep, diet, memory surveys) will be performed pre- and post-exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or above
* Enrollment in Stay Strong Stay Healthy Program
* Strength training < 2 hours/week for past 3 months

Exclusion Criteria:

* Not enrolled in Stay Strong Stay Healthy Program
* Strength training > 2 hours/week for past 3 months
* Donated more than 463 ml of blood in past 8 weeks
* Physician discouraged to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Muscle electrical activity | Change in muscle electrical activity in 8 weeks in response to resistance exercise program
  Measurement of muscle electrical activity is made using electromyography technique at baseline and after 8 weeks of resistance exercise.

SECONDARY OUTCOMES:
Exert muscle power/strength | Change in muscle power/strength in 8 weeks in response to resistance exercise program
  Measurement of muscle power/strength is made using hand dynamometer at baseline and after 8 weeks of resistance exercise.
Muscle mass loss | Change in muscle mass in 8 weeks in response to resistance exercise program
  Changes in the muscle mass is made using dual x-ray absorptiometry technique at baseline and after 8 weeks of resistance exercise.
Ability to think or remember | Changes in thinking and cognitive abilities in 8 weeks in response to resistance exercise program
  Changes in ability to think or remember is measured by using standard survey (Self Administered Gerocognitive Exam Form -1) at baseline and after 8 weeks of resistance exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Ball, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geirsdottir OG, Arnarson A, Briem K, Ramel A, Jonsson PV, Thorsdottir I. Effect of 12-week resistance exercise program on body composition, muscle strength, physical function, and glucose metabolism in healthy, insulin-resistant, and diabetic elderly Icelanders. J Gerontol A Biol Sci Med Sci. 2012 Nov;67(11):1259-65. doi: 10.1093/gerona/gls096. Epub 2012 Apr 10. PMID 22496538
- [Background] Sale DG. Neural adaptation to resistance training. Med Sci Sports Exerc. 1988 Oct;20(5 Suppl):S135-45. doi: 10.1249/00005768-198810001-00009. PMID 3057313
- [Background] Pollock ML, Franklin BA, Balady GJ, Chaitman BL, Fleg JL, Fletcher B, Limacher M, Pina IL, Stein RA, Williams M, Bazzarre T. AHA Science Advisory. Resistance exercise in individuals with and without cardiovascular disease: benefits, rationale, safety, and prescription: An advisory from the Committee on Exercise, Rehabilitation, and Prevention, Council on Clinical Cardiology, American Heart Association; Position paper endorsed by the American College of Sports Medicine. Circulation. 2000 Feb 22;101(7):828-33. doi: 10.1161/01.cir.101.7.828. No abstract available. PMID 10683360
- [Background] Mayer F, Scharhag-Rosenberger F, Carlsohn A, Cassel M, Muller S, Scharhag J. The intensity and effects of strength training in the elderly. Dtsch Arztebl Int. 2011 May;108(21):359-64. doi: 10.3238/arztebl.2011.0359. Epub 2011 May 27. PMID 21691559
- [Background] Kraemer WJ, Ratamess NA. Hormonal responses and adaptations to resistance exercise and training. Sports Med. 2005;35(4):339-61. doi: 10.2165/00007256-200535040-00004. PMID 15831061
- [Background] Macaluso A, De Vito G. Muscle strength, power and adaptations to resistance training in older people. Eur J Appl Physiol. 2004 Apr;91(4):450-72. doi: 10.1007/s00421-003-0991-3. Epub 2003 Nov 25. PMID 14639481
- [Result] Ball S, Gammon R, Kelly PJ, Cheng AL, Chertoff K, Kaume L, Abreu EL, Brotto M. Outcomes of Stay Strong, Stay Healthy in community settings. J Aging Health. 2013 Dec;25(8):1388-97. doi: 10.1177/0898264313507318. Epub 2013 Oct 22. PMID 24150062